CLINICAL TRIAL: NCT05829343
Title: RObotic Vs LAparoscopic Colectomy for DIverticulitis. a Multicenter Observational Prospective Study.
Brief Title: RObotic Versus LAparoscopic Colectomy for DIverticulitis.
Acronym: ROLADI
Status: Recruiting | Type: Observational
Sponsor: S.M. Misericordia Hospital (Other)
Responsible Party: Principal Investigator, Giuliani Giuseppe, MD - Assistant surgeon, S.M. Misericordia Hospital
Other Study IDs: ROLADI - 1.0
Record Dates: First submitted 2023-04-11; First posted 2023-04-25 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Diverticular Diseases; Diverticulitis
Keywords: Diverticular Disease; Robotic surgery; Laparoscopic surgery; Minimal invasive surgery; Colorectal surgery
MeSH Terms: conditions — Diverticular Diseases; Diverticulitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Robotic surgery group: Patients with diverticular disease resected with a robotic approach.
  Interventions: Procedure: Robotic left colectomy
- Laparoscopic surgery group: Patients with diverticular disease resected with a laparoscopic approach.
  Interventions: Procedure: Laparoscopic Left colectomy

INTERVENTIONS:
Procedure: Laparoscopic Left colectomy — Patients are treated with a laparoscopic approach as the standard of care for the treatment of left-sided colonic diverticular disease, depending on the experience of the surgeon or institution.
  Groups: Laparoscopic surgery group
Procedure: Robotic left colectomy — Patients are treated with a robotic approach as the standard of care for the treatment of left-sided colonic diverticular disease, depending on the experience of the surgeon or institution.
  Groups: Robotic surgery group

SUMMARY:
Over the last decade there has been a growing interest toward the application of robotic approach for diverticular disease. The evidence available on the literature showed that robotic approach, compared to the laparoscopic surgery, offers significant advantages in terms of conversion rate and shortened hospital stay for the treatment of diverticular disease.

The investigators aimed at evaluating whether robotic colectomy may offer some advantages over the laparoscopic approach for surgical treatment of diverticular disease by analyzing a one year multicenter prospective study.

Primary objective is to evaluate if robotic approach reduce the rate of conversion to open approach compared to laparoscopic surgery. Secondary objective is to assess difference between the two approaches in terms of rate of intraoperative complication, postoperative morbidities (according with Clavien and Dindo Classification), hospital stay and at one year follow up. Inclusion criteria are: elective colectomy for complicated or non-complicated diverticular disease performed with laparoscopic or robotic approach and age between 18 and 90 years. Exclusion criteria are non-elective colectomy (emergency resection), open procedure, diverticular resection performed during other procedure (i.e. colectomy for cancer). Data will be collected in one year from the start of the study.

Due to the lack of available evidence, it is impossible to draw definitive conclusions. With this study, the investigators hope to clarify the role of the robotic approach in the treatment of diverticular disease.

DETAILED DESCRIPTION:
Background Over the past decade, there has been a growing interest in the use of robotic surgery for diverticular disease (DD). The evidence available in the literature is based on retrospective studies and two meta-analyses1,2. To date, the robotic approach offers significant advantages over laparoscopic surgery in terms of conversion rate and shortened hospital stay for the treatment of diverticular disease.

The investigators aimed to evaluate whether elective robotic colectomy may offer some advantages over the laparoscopic approach for surgical treatment of diverticular disease performing a prospective multicenter study.

Methods and Materials This is a multi-center, prospective, not-for-profit cohort study that will enroll patients undergoing elective or delayed urgent surgical treatment for left-sided colonic diverticular disease. The enrollment period will be one year, followed by one year of follow-up. The study will start in Juin 2023.

Data will be collected in a prospective database using an easy to fill out Google form, also available on mobile devices.

Several preoperative, intraoperative and postoperative outcomes will be analyzed.

OUTCOMES Pre-Operative

* Demographic Outcomes: Age, gender, body mass index (BMI), American Society of Anesthesiologists (ASA), Charlson Comorbidity Index (CSI: https://www.mdcalc.com/calc/3917/charlson-comorbidity-index-cci)
* Indications for surgery:
* Complicated DD: colonic stenosis, abscess, fistula, others;
* Recurrent DD: multiple episodes of diverticulitis affecting quality of life;
* Planned vascular ligation (inferior mesenteric artery vs. sigmoid arteries)
* Preoperative bowel preparation
* Indication for minimally invasive approach pursued (Why Rob vs Lap)

Intraoperative

* Surgical approach (laparoscopic or robotic)
* Intraoperative findings (sigmoid stenosis, stricture, adhesion, fistula)
* Intraoperative complications (specify types)
* Conversion to open approach
* Operative times
* Effective vessel ligation
* Splenic flexure mobilization
* Type of colon resection (sigmoidectomy, left colectomy, anterior rectal resection, Hartmann procedure)
* Stoma (ileostomy vs. colostomy)
* Associated procedures
* Specimen extraction (midline, off midline, suprapubic or natural orifice) Postoperative
* 30-day postoperative complications (Clavien-Dindo classification)
* 30-day reoperation
* 30-day readmission
* Length of stay LOS
* Time to return to work (days)
* 30 days - Mortality
* One-year follow-up

Sample size The estimated sample sizes for the study using a proportion of 0.125 for Laparoscopic approach and a proportion of 0.074 for Robotic approach, and a risk of conversion rate OR=0.56 (IC95% 0.45-0.70), is at least 1450 patients (725 for the group - alpha = 0.0500, power = 0.9000, delta = 0.5600). MICE (Multivariate Imputation via Chained Equations) is the procedure used to impute missing data for explanatory variables. In this approach, instead of imputing all missing values with a single value (mean/median), the statistical information is derived from the median), it takes into account the statistical information derived from the distribution of the other variables. The missing values are considered as an outcome to be predicted. This allows to take into account the correct variability in the entire data set and to obtain estimates that are as unbiased as possible.

Statistical Analysis The quantitative variables included in the study are expressed as mean ± standard deviation, median and range (distance between maximum and minimum values), both at the overall level and by surgical approach. The qualitative (categorical) variables are presented as percentages and absolute values, both at a general level and divided by surgical approach. It will be evaluated, if necessary, to perform a propensity score matching procedure between the two approaches (Rob and Lap), using the nearest neighbor matching technique, without replacement. Demographics, pre-operative and intra-operative characteristics are used in the propensity score logistic regression models to minimize selection bias, by assembling a matched cohort in which confounding factors are balanced between the two groups. In the matched cohort bivariate analyses are performed to .compare the primary and secondary outcomes between the two groups.

The comparison between the quantitative variables of interest is performed by the two-tailed Student T-test (in case of heteroskedasticity of variances) or with nonparametric tests, such as the Mann-Whitney U test or theKruskal-Wallis test. The comparison between qualitative variables of interest is carried out to evaluate the association or not between them, through an extension of the chi-square test suitable for multicenter studies (the Cochran - Mantel - Haenszel test).

For the entire cohort multivariate logistic regression models are performed to test the effect of surgical approach on primary and secondary outcomes.

Ethics and dissemination The trial will be conducted in accordance with the Declaration of Helsinki and in compliance with the Good Clinical Practice, Principle E6 (R2). The study will be approved by the Ethics Committee of the coordinating center (Comitato Etico di Area Vasta Sud Est Dipartimento Politiche del Farmaco e Attività Farmaceutiche Segreteria Amministrativa) and then will be registered at ClinicalTrial.gov. Subsequently, all participating centers will receive approval to participate from the local institutional review board. Authorship for written publications will be confirmed for all participating investigators (2 investigators per center). Anonymized participant-level data sets will be made available upon reasonable upon reasonable request by contacting the principal investigator. Study results will be presented at international or national meetings and published in surgical journals.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Elective or delayed urgency colorectal resection for left-sided DD
* Fully minimally invasive (robotic or laparoscopic) procedures.

Exclusion Criteria:

* Age < 18 years
* Urgent resection for DD
* Hybrid minimally invasive resection
* Conventional open resection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diverticular disease of the left colon with surgical indication.
Sampling Method: Non-Probability Sample
Enrollment: 1450 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Conversion rate | One year
  The primary objective is to evaluate whether the robotic approach reduces the rate of conversion to open surgery compared to laparoscopic surgery.

SECONDARY OUTCOMES:
Intra - operative complications | One year
  The first secondary outcome measure is to assess the difference between the two approaches in terms of intra-operative complications (e.g. bleeding, spleen injury, ureteral injury, bowel perforation)
Operative time | One year
  Evaluate the possible difference in terms of operative time (expressed in minutes) between the two groups, to assess whether the robotic approach has a longer operative time than the laparoscopic approach.
Complicated disease | One year
  Evaluate the difference between the two approaches in the number of complicated cases performed. For example, analyze whether one group performs more complicated diverticular disease (e.g., colonic stenosis, colorectal fistula, intraperitoneal abscess) than the other.
30 day Post - operative complications | One year
  Another secondary outcome measure is to assess the difference between the two groups in terms of post-operative complications (using the Clavien and Dindo classification).
30-day Post - operative re-operation | One year
  Evaluate the possible difference in term of rate of re-operation between the two groups within 30 day after surgery.
30-day Post - operative mortality | One year
  Evaluate the possible difference in term of rate of mortality between the two groups within 30 day after surgery.
Length of hospital stay | One year
  Evaluate the possible difference in term of length of hospital stay (expressed in day) between the two groups.
Time to return at work | One year
  Evaluate the possible difference in time to return to work (expressed in days from surgery) between the two groups.
One year follow up | Two years
  Evaluate the possible difference in terms of disease recurrence or incisional hernia, between the two groups at one year after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of General and Emergency Surgery. Misericordia Hospital. Director: Coratti Andrea, MD, Grosseto, Tuscany, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Giuliani G, Guerra F, Coletta D, Giuliani A, Salvischiani L, Tribuzi A, Caravaglios G, Genovese A, Coratti A. Robotic versus conventional laparoscopic technique for the treatment of left-sided colonic diverticular disease: a systematic review with meta-analysis. Int J Colorectal Dis. 2022 Jan;37(1):101-109. doi: 10.1007/s00384-021-04038-x. Epub 2021 Oct 1. PMID 34599362
- [Background] Larkins K, Mohan H, Apte SS, Chen V, Rajkomar A, Larach JT, Smart P, Heriot A, Warrier S. A systematic review and meta-analysis of robotic resections for diverticular disease. Colorectal Dis. 2022 Oct;24(10):1105-1116. doi: 10.1111/codi.16227. Epub 2022 Aug 9. PMID 35723895